CLINICAL TRIAL: NCT01354301
Title: Efficacy and Safety of Induction Strategies Combined With Low Tacrolimus Exposure in Kidney Transplant Recipients Receiving Everolimus or Sodium Mycophenolate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Helio Tedesco Silva Junior, PhD, Hospital do Rim e Hipertensão
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ABR18T
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Cytomegalovirus Infection; Renal Transplant Failure; Transplant; Complication, Rejection
Keywords: kidney transplantation; thymoglobulin; everolimus
MeSH Terms: conditions — Cytomegalovirus Infections; Rejection, Psychology | interventions — thymoglobulin; Everolimus; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Thymoglobulin and everolimus (Experimental): single dose antithymocyte globulin, reduced concentration tacrolimus, everolimus starting at day 2 posttransplant and prednisone
  Interventions: Drug: Thymoglobulin; Drug: Everolimus; Drug: Tacrolimus
- Basiliximabe and everolimus (Experimental): basiliximab, reduced concentration tacrolimus, everolimus starting at day 2 posttransplant and prednisone
  Interventions: Drug: Everolimus; Drug: Basiliximabe; Drug: Tacrolimus
- Basiliximabe and mycophenolate (Active Comparator): basiliximab, reduced concentration tacrolimus, mycophenolate and prednisone.
  Interventions: Drug: Basiliximabe; Drug: mycophenolate sodium; Drug: Tacrolimus

INTERVENTIONS:
Drug: Thymoglobulin — intravenously, beginning within the first 24 hours after graft revascularization. Pre-treatment includes hydrocortisone and dipyrone before antithymocyte globulin infusion, which will be reconstituted according to the package insert.
  Arms: Thymoglobulin and everolimus
Drug: Everolimus — initial 0.75 mg BID dose of everolimus on day 2. Doses will be adjusted from day 5 on to maintain everolimus whole blood trough concentrations between 4-8 ng/ml.
  Arms: Basiliximabe and everolimus; Thymoglobulin and everolimus
Drug: Basiliximabe — days 0 and 4, according to the package insert instructions.
  Arms: Basiliximabe and everolimus; Basiliximabe and mycophenolate
Drug: mycophenolate sodium — 720 mg BID. This dose will be reduced according to adverse events.
  Arms: Basiliximabe and mycophenolate
Drug: Tacrolimus — 0.05 mg/kg BID beginning on day 1. Doses will be adjusted to maintain tacrolimus whole blood trough concentrations between 3-5 ng/ml.
  Arms: Thymoglobulin and everolimus
Drug: Tacrolimus — 0.1 mg/kg BID beginning on day 1. Doses will be adjusted to maintain tacrolimus whole blood trough concentrations between 3-8 ng/ml and 3-5 ng/ml after 3 months.
  Arms: Basiliximabe and everolimus
Drug: Tacrolimus — 0.1 mg/kg BID beginning on day 1. Doses will be adjusted to maintain tacrolimus whole blood trough concentrations between 3-8 ng/ml.
  Arms: Basiliximabe and mycophenolate

SUMMARY:
Despite the improvement of efficacy results with current immunosuppressive regimens (about 15% of incidence of acute rejection), the security schemes used do not show the same results.The most worldwide used regime is tacrolimus, mycophenolate and prednisone. Despite the favorable efficacy results in our population, the use of this combination is associated with higher incidence of viral infections such as cytomegalovirus, and gastrointestinal events, two common causes of hospital readmissions after renal transplantation at our institution.Given this, the investigators propose a study of our own initiative that attends our local needs: identify the best strategy among the therapeutic options available to maintain the result of current effectiveness and improve the safety profile for kidney transplant recipients.This protocol is a prospective, randomized, single center, designed to compare the safety and efficacy of three immunosuppressive regimens: (1) single dose of antithymocyte globulin, reduced exposure to tacrolimus, everolimus starting on day 2 after transplantation and prednisone; ( 2) basiliximab, reduced exposure to tacrolimus, everolimus starting on day 2 after transplantation and prednisone; (3-control group) basiliximab, reduced exposure to tacrolimus, mycophenolate and prednisone.Our hypothesis is that a single dose of antithymocyte globulin or basiliximab induction therapy in combination with low doses of tacrolimus, everolimus and prednisone results in comparable efficacy observed in patients receiving tacrolimus / mycophenolate / prednisone, but with a better safety profile.

To ensure efficacy, the investigators added to the regimes the induction with monoclonal or polyclonal antibody. To improve the toxicities associated with the current scheme, the investigators replace the use of mycophenolate by everolimus and the investigators reduced the dose of tacrolimus.

Patients will be monitored for blood levels of tacrolimus and everolimus to ensure adequate exposure to immunosuppressive agents.

DETAILED DESCRIPTION:
Primary end-point: The incidence of CMV infection or disease during the first year of transplantation.Secondary main end-point: the incidence of treatment failure defined as a composite end-point of BCAR, graft loss, death, loss to follow up.

The investigators anticipate enrolling 300 patients within 12 months. Only low risk adult candidates for first renal transplants from living or deceased donors will be considered for enrollment. Patients will be excluded if they have been receiving immunosuppressive therapy before transplantation; have received an investigational medication within the past 30 days; have a known contraindication to the administration of antithymocyte globulin; if tested positive for human immunodeficiency virus (HIV); if had had cancer (except nonmelanoma skin cancer) within the previous 2 years. Pregnant women, nursing mothers, and women of childbearing potential who will be not using condoms or oral contraceptives will be excluded. Patients with any panel reactive antibody (PRA) equal to or above 50%, class I or class II, will also be excluded. Study visits will be performed at pre transplant, days 0, 1, 7, every week up to month 6 and month 12.

ELIGIBILITY:
Inclusion Criteria:

* low risk adult candidates for first renal transplants from living or deceased donors

Exclusion Criteria:

* receiving immunosuppressive therapy before transplantation;
* have received an investigational medication within the past 30 days;
* have a known contraindication to the administration of antithymocyte globulin;
* tested positive for human immunodeficiency virus (HIV);
* had had cancer (except nonmelanoma skin cancer) within the previous 2 years;
* Pregnant women, nursing mothers, and women of childbearing potential who will be not using condoms or oral contraceptives will be excluded;
* Patients with any panel reactive antibody (PRA) equal to or above 50%, class I or class II.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
incidence of CMV infection or disease | 1 year

SECONDARY OUTCOMES:
incidence of treatment failure defined as a composite end-point of BCAR, graft loss, death, loss to follow up. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hélio Tedesco, MD, Principal Investigator — Hospital do Rim e Hipertensão - Fundação Oswaldo Ramos
Locations (1):
- Hospital do rim e Hipertensao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Nunes Ficher K, Dreige Y, Gessolo Lins PR, Nicolau Ferreira A, Toniato de Rezende Freschi J, Linhares K, Stopa Martins S, Custodio L, Cristelli M, Viana L, Wagner Santos D, de Marco R, Gerbase-DeLima M, Proenca H, Aguiar W, Nakamura M, Rosso Felipe C, Medina Pestana J, Tedesco Silva H Jr. Long-term Efficacy and Safety of Everolimus Versus Mycophenolate in Kidney Transplant Recipients Receiving Tacrolimus. Transplantation. 2022 Feb 1;106(2):381-390. doi: 10.1097/TP.0000000000003714. PMID 33988338
- [Derived] Tedesco-Silva H, Felipe C, Ferreira A, Cristelli M, Oliveira N, Sandes-Freitas T, Aguiar W, Campos E, Gerbase-DeLima M, Franco M, Medina-Pestana J. Reduced Incidence of Cytomegalovirus Infection in Kidney Transplant Recipients Receiving Everolimus and Reduced Tacrolimus Doses. Am J Transplant. 2015 Oct;15(10):2655-64. doi: 10.1111/ajt.13327. Epub 2015 May 18. PMID 25988935